CLINICAL TRIAL: NCT06190327
Title: Effects of a Blended Indoor and Outdoor Physical Exercise Program on Depressive Symptoms in Hong Kong Older Adults: a Randomized Controlled Trial
Brief Title: Effects of a Blended Indoor and Outdoor Physical Exercise Program on Depressive Symptoms in Hong Kong Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05200098
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Depressive Symptoms
Keywords: depressive symptoms; older adults; multicomponent structured exercise; blended indoor and outdoor environment; indoor exercise; connectedness to nature
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: This study follows a randomized controlled experimental design (RCT), parallel type with three groups and being assessed in a pretest, posttest, and after three months of the completion of the intervention. The participants will be randomly allocated to two experimental group, and one non-exercise control group. The non-exercise control group continue to maintain their daily routine and keep diaries to record . To monitor the control condition, participants will need to keep diaries to record their daily physical exercise, medicines used, illness and participation in other health-related activities. The research assistant will give telephone calls to the participants biweekly to check their diaries and identify if they change their lifestyles or experience adverse events. Two exercise groups, one group will perform multicomponent structured exercise in blended indoor and outdoor setting, the other group will conduct the same exercise only in indoor setting.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- blended indoor and outdoor multicomponent structured exercise group (Experimental): Participants will receive a 16-week blended indoor and outdoor multicomponent structured exercise program, with 2 sessions per week (90 mins/session).
  Interventions: Behavioral: Blended indoor and outdoor multicomponent structured exercise
- indoor-only multicomponent structured exercise group (Active Comparator): Participants will receive a 16-week indoor-only multicomponent structured exercise program, with 2 sessions per week (90 mins/session).
  Interventions: Behavioral: Indoor-only multicomponent structured exercise
- control group (No Intervention): The control group will not receive any intervention during the whole project.

INTERVENTIONS:
Behavioral: Blended indoor and outdoor multicomponent structured exercise — Participants will receive a 16-week blended indoor and outdoor multicomponent structured exercise program, with 2 sessions per week (90 mins/session). Session 1/week will conduct in indoor setting, while session 2/week will conducted in outdoor setting (park). Each session will comprise 10-min warm-up, 30-min aerobic training, 20-min muscle strength, 20-min postural balance training, and 10-min cool-down.
  Arms: blended indoor and outdoor multicomponent structured exercise group
Behavioral: Indoor-only multicomponent structured exercise — Participants will receive a 16-week indoor-only multicomponent structured exercise program, with 2 sessions per week (90 mins/session). Both two sessions will conducted in indoor setting. Each session will comprise 10-min warm-up, 30-min aerobic training, 20-min muscle strength, 20-min postural balance training, and 10-min cool-down.
  Arms: indoor-only multicomponent structured exercise group

SUMMARY:
Depression is a mental health problem often occurring in the elderly. Performing physical exercise is a key element in decreasing depressive symptoms in older adults. Most studies investigating depression and physical exercise have focused on structured exercise comprise of one or two exercise components and based on the clinical patients associated with major depression. There is limited research combining multicomponent (aerobic+resistance+balance) in an exercise program and targeting non-clinical adults with depressive symptoms, with even less available for older adults.

More attention has been paid to the role of outdoor exercise on human health. Exercise in a natural environment may provide greater physiological and psychological benefits compared to indoor exercise. Findings demonstrated that green exercise provides double the beneficial effect on improving depression among adults. Although green exercise shows effects on the improvement of depression, recently a review has indicated that structured exercise programs in older adults with depressive symptoms were mainly conducted in the indoor environment. Compared with outdoor exercise which is easily influenced by the weather and with low access of available facilities, indoor exercise is more comfortable, quiet, and convenient to operate especially for older adults. Considering the high relevance between nature and mental health, the combination of indoor and outdoor exercise programs might be able to maximize intervention effectiveness while maintaining the benefits for each type of intervention.Therefore, more rigorous RCT studies in this field are needed, particularly for non-clinical older adults with depressive symptoms.

DETAILED DESCRIPTION:
The 16-week double-blinded RCT (2 sessions/week, 90 min/session) will include community-dwelling older adults aged 60 to 74 years old with depressive symptoms. Participants will be randomized to one of three groups (a blended indoor and outdoor group, an indoor-only group or a control group) using 1:1:1 allocation ratio. Structured exercise training with multicomponent (aerobic, muscle strength, balance) will be conducted in two intervention groups. The intervention effects will be evaluated on depressive symptoms, physical fitness, physical activity enjoyment and connectedness to nature. All measured data will be collected at the pre-intervention, post-intervention, and 3-month follow up stages.

ELIGIBILITY:
Inclusion Criteria:

* 60 to 74 years at the start date of the project.
* Chinese version of Geriatric Depression Scale (GDS-C) scoring 5-15 (i.e., mild to serve level of depressive symptoms).
* Passing the PAR-Q plus screening or with the physician's approval for readiness to participate in high-intensity exercise.

Exclusion Criteria:

* Having cognition impairment regarded by specialists.
* are attending other health projects related to physical exercise.

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-11-03 (Estimated)

PRIMARY OUTCOMES:
Self-reported depressive symptoms | Outcome evaluations will be performed three times at pre-intervention (T1 baseline), after 16-weeks intervention (T2 post-test), and 3 months after intervention completion (T3 follow-up test).
  The Chinese version of the 15-item Geriatric Depression Scale (GDS-C) will be used to measure the subjective depression level. The GDS are the most widely used scales for the detection of depression symptoms in older adults (Cronbach's α = .81 -.83).
Concentration of saliva cortisol | Evaluations of concentration of saliva cortisol will be performed three times at pre-intervention (T1 baseline), after 16-weeks intervention (T2 post-test), and 3 months after intervention completion (T3 follow-up test).
  Objective biomarker of depression will be measured in salivary cortisol. All participants will be provided with three salivette tubes and be asked to collect the saliva samples (2-3 ml) at awakening and 30 mins after awakening, respectively. All saliva samples for all subjects will be collected at the same time of day and samples will not be taken on days in which participants are sick with a fever. The salivette tubes will be stored in the freezer zone until to be tested. ELISA KIT protocol will be used to be followed to collect and analyze the samples in each assessment.

SECONDARY OUTCOMES:
Physical fitness | Outcome evaluations will be performed three times at pre-intervention (T1 baseline), after 16-weeks intervention (T2 post-test), and 3 months after intervention completion (T3 follow-up test).
  Physical fitness will be assessed using the Senior Fitness Test (SFT) battery. There are seven testing items measuring all five dimensions, including the body mass index (BMI), 30s chair stand for lower limbs' muscle strength, 30s arm curl for upper limbs' muscle strength, 2-min step test for aerobic endurance, chair sit-and-reach test for lower body flexibility, back scratch test for upper body flexibility, and 8ft up-and-go test for mobility and dynamic balance.
Loneliness | Evaluations of concentration of saliva cortisol will be performed three times at pre-intervention (T1 baseline), after 16-weeks intervention (T2 post-test), and 3 months after intervention completion (T3 follow-up test).
  The 6-item De Jong Gierveld Loneliness Scale with Chinese version will be applied for assessing loneliness. This scale has been shown a sound reliability and validity for older adults in Hong Kong (Cronbach's alpha=0.76). Item 1 to item 3 as negatively worded items will be measured "emotional loneliness", answer "yes" will score 1, answer "more or less" will score 1, answer "no" will score 0. Item 4 to item 6 as positively worded items will be used to assessed "social loneliness", answer "yes" will score 0, answer "more or less" will score 1, answer "no" will score 1.
Physical activity enjoyment | Evaluations of concentration of saliva cortisol will be performed three times at pre-intervention (T1 baseline), after 16-weeks intervention (T2 post-test), and 3 months after intervention completion (T3 follow-up test).
  The Chinese version of the 8-item physical activity enjoyment scale (PACES) will be measured participant's enjoyment level after engaging in blended indoor and outdoor multicomponent exercise program. This scale has revealed strong internal consistency and reliability among Hong Kong older adults (Cronbach's alpha=0.92). It will be scored by 7 bipolar rating, from one extreme to the other extreme, for example, from "it's very pleasant" to "it's very unpleasant".
Connectedness to nature | Evaluations of concentration of saliva cortisol will be performed three times at pre-intervention (T1 baseline), after 16-weeks intervention (T2 post-test), and 3 months after intervention completion (T3 follow-up test).
  The 14-item connectedness to nature scale (CNS) with Chinese version will be used to measure the sense of belonging to the natural world. This five-point scale, ranging from 1 "strongly disagree" to 5 "strongly agree".

OTHER OUTCOMES:
Self-reported Rate of Perceived Exertion (RPE) | RPE will be asked at the end of main exercise at each exercise session during the 16-weeks intervention.
  Older adults will be asked about the self-reported Rate of Perceived Exertion (RPE Borg CR-10 category scale) after they complete the main exercise training in each session.
Process evaluation of intervention program | Outcome evaluations will be conducted at the completion of 16-weeks intervention.
  A process evaluation scale of the intervention process will be developed for this study based on the previous framework of process evaluation for the intervention study. This scale with 10 items using a 5-point (strongly unsatisfied, unsatisfied, neutral, satisfied, and strongly satisfied). The score on this scale ranges from 10 to 50, a higher score shows higher satisfaction with the intervention program.

CONTACTS AND LOCATIONS:
Overall Officials: Yanping Duan, P.hD, Principal Investigator — Hong Kong Baptist Univeristy; Department of Sport, Physical Education and Health
Locations (1):
- Bliss District Elderly Community Centre, Kowloon Bay, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wei J, Hou R, Zhang X, Xu H, Xie L, Chandrasekar EK, Ying M, Goodman M. The association of late-life depression with all-cause and cardiovascular mortality among community-dwelling older adults: systematic review and meta-analysis. Br J Psychiatry. 2019 Aug;215(2):449-455. doi: 10.1192/bjp.2019.74. Epub 2019 Apr 10. PMID 30968781
- [Background] Cheung KCK, Chou KL. Poverty, deprivation, and depressive symptoms among older adults in Hong Kong. Aging Ment Health. 2019 Jan;23(1):22-29. doi: 10.1080/13607863.2017.1394438. Epub 2017 Oct 31. PMID 29086588
- [Background] Zhao SZ, Wong JYH, Luk TT, Wai AKC, Lam TH, Wang MP. Mental health crisis under COVID-19 pandemic in Hong Kong, China. Int J Infect Dis. 2020 Nov;100:431-433. doi: 10.1016/j.ijid.2020.09.030. Epub 2020 Sep 16. PMID 32947051
- [Background] Teychenne M, Ball K, Salmon J. Sedentary behavior and depression among adults: a review. Int J Behav Med. 2010 Dec;17(4):246-54. doi: 10.1007/s12529-010-9075-z. PMID 20174982
- [Background] Catalan-Matamoros D, Gomez-Conesa A, Stubbs B, Vancampfort D. Exercise improves depressive symptoms in older adults: An umbrella review of systematic reviews and meta-analyses. Psychiatry Res. 2016 Oct 30;244:202-9. doi: 10.1016/j.psychres.2016.07.028. Epub 2016 Jul 22. PMID 27494042
- [Background] Eigenschenk B, Thomann A, McClure M, Davies L, Gregory M, Dettweiler U, Ingles E. Benefits of Outdoor Sports for Society. A Systematic Literature Review and Reflections on Evidence. Int J Environ Res Public Health. 2019 Mar 15;16(6):937. doi: 10.3390/ijerph16060937. PMID 30875938
- [Background] Askari J, Saberi-Kakhki A, Yassini SM. The Effect of Aerobic Indoor Exercise Compared with Green Exercise on Different Symptoms of Depression: An Investigation of Psychological Mediators of Stress and Coping. Open Journal of Medical Psychology. 2017 Jul 3;6(03):197.
- [Background] Li N, Wu J. Revise of the Connectedness to Nature Scale and its Reliability and Validity. China Journal of Health Psychology. 2016 Mar 22;24(9):1347-50.
- [Background] Loureiro A, Veloso TJ. Outdoor exercise, well-being and connectedness to nature. Psico. 2014 Mar;45(3):299-304.
- [Background] Cheng ST, Chan AC. A brief version of the geriatric depression scale for the chinese. Psychol Assess. 2004 Jun;16(2):182-6. doi: 10.1037/1040-3590.16.2.182. PMID 15222814
- [Background] Chiu HF, Lee H, Chung W, Kwong P. Reliability and validity of the Cantonese version of mini-mental state examination-a preliminary study. Hong Kong Journal of Psychiatry. 1994;4(2):25.
- [Background] Chung PK, Zhao YN, Quach, B, Liu JD. The Use of the Cantonese Rating of Perceived Exertion Scale in Older People. Proceedings of the 12th SCSEPF Annual Conference. 2013.
- [Background] Chung PK, Leung KM. Psychometric Properties of Eight-Item Physical Activity Enjoyment Scale in a Chinese Population. J Aging Phys Act. 2018 Oct 12:1-6. doi: 10.1123/japa.2017-0212. Online ahead of print. PMID 29722637
- [Derived] Cheng S, Duan Y, Lau WB, Liang W, Chan NJ, Young KD, Baker JS, Lau TJ. Effect of a blended indoor and outdoor multicomponent structured exercise on depressive symptoms in Hong Kong older adults: study protocol of a randomized controlled trial. BMC Public Health. 2025 Nov 14;25(1):3949. doi: 10.1186/s12889-025-25244-0. PMID 41239372